CLINICAL TRIAL: NCT02085356
Title: Implementing Comprehensive PMTCT and HIV Prevention for South African Couples
Brief Title: Implementing a Comprehensive Prevention of Mother-to-Child Transmission of HIV Program for South African Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Human Sciences Research Council (Other Government)
Responsible Party: Principal Investigator, DEBORAH JONES, Research Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20130238; 1R01HD078187 (NIH)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: HIV; Pregnancy
Keywords: HIV; PMTCT; South Africa; Couples; Male involvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention women with partners (Experimental): Women will enroll with male partners and both members of the couple will attend the Protect your Family intervention
  Interventions: Behavioral: Protect your family
- Intervention women without partners (Experimental): Women will enroll alone and will attend the Protect your Family Intervention without a partner
  Interventions: Behavioral: Protect your family
- Control women with partners (No Intervention): Women will enroll with male partners and both members of the couple will attend time-matched video sessions
- Control women alone (No Intervention): Women will enroll alone and will attend time-matched video sessions

INTERVENTIONS:
Behavioral: Protect your family — "Protect Your Family" intervention is a manualized, closed, structured behavioral risk reduction program targeting HIV, stigma, disclosure, communication, intimate partner violence (IPV), PMTCT knowledge, safer conception, family planning and dual method sexual barrier use.
  Intervention participants will attend 3 prenatal weekly 2 hour gender-specific (male or female, 5-7 participants) group sessions followed by 1 individual counseling session and 2 monthly couples or individual (women-only) counseling sessions (1 prenatal, 2 postpartum) led by study-trained clinic staff (e.g., nurses, HIV counseling and testing (HCT) counselors) plus standard of care (PMTCT)
  Arms: Intervention women with partners; Intervention women without partners

SUMMARY:
This study will test the effectiveness of a behavioral intervention to increase Prevention of Mother-to-Child Transmission of HIV (PMTCT) protocol uptake among South African HIV positive pregnant women. This study will also determine whether the participation of male partners will have additional positive impact on PMTCT uptake. The intervention will utilize a combination of both gender-concordant groups and individual or couples counseling strategies, before and after birth. During antenatal care, the intervention will use a gender-concordant group format to address PMTCT information, HIV disclosure, coping with stigma, intimate partner violence, and adherence to the overall PMTCT protocol. Just prior to birth and following birth, the intervention will shift to individual or couples-based counseling, targeting medication adherence, safer infant feeding, and family planning. It is hypothesized that women attending the intervention will be more likely to properly take HIV medication before birth and provide it to their infants. Additionally, it is hypothesized that male partner involvement will further increase the likelihood that mothers will take their HIV medication as prescribed and provide it to their infants.

DETAILED DESCRIPTION:
Abstract. In rural South Africa, only two-thirds of HIV+ pregnant women seeking antenatal care at community health centers took full advantage of available "prevention of mother-to-child transmission" (PMTCT) services in 2010 (SADOH). While engagement of male partners has been encouraged as a potential means of increasing PMTCT uptake, men have been reluctant to accompany their wives/partners to antenatal care.

Recent studies generally support male involvement in promoting PMTCT, but the nature and impact of that involvement is unclear and untested. It is also clear that factors such as stigma, disclosure and intimate partner violence pose significant barriers to PMTCT uptake and retention in care, suggesting that male involvement may be "necessary, but not sufficient" to accomplish the WHO goal of <5% infant HIV incidence. Additional measures may be needed to increase participation by HIV positive pregnant women in PMTCT.

In 2011, Mpumalanga Province had the highest rates of HIV in the country (36.7%) and rates of infant HIV incidence in rural clinics ranged up to 50%. Rates of PMTCT uptake in the Province have been among the lowest in South Africa (69%). This application proposes to expand on a successful PEPFAR- supported, PMTCT couples intervention pilot study conducted in Mpumalanga Province, ("Vikela Umndeni: Protect Your Family") to include a more representative population of HIV positive pregnant women and their partners, the primary objective being to determine whether male partner involvement plus a behavioral intervention would significantly reduce infant HIV incidence by increasing levels of adherence to ARV/ PMTCT protocols, including breastfeeding and family planning, during the antenatal and post-natal periods.

The proposed study will enroll two cohorts of HIV positive pregnant women recruited from 12 randomly assigned Community Health Centers (6 experimental, 6 control): a) Women attending without their male partners (n = 720), followed by b) Women attending with their male partners (n = 720 couples), to determine whether the influence of male participation itself or combined with a behavioral PMTCT intervention can significantly reduce infant HIV infection ante-, peri- and post-natally. It is our intention to significantly increase PMTCT participation from current levels (69%) in Mpumalanga Province to 90-95% through engaging women and couples in a unique, controlled, six session ante- and post-natal risk-reducing/PMTCT promotion intervention addressing the barriers to PMTCT (e.g., stigma, disclosure, intimate partner violence, communication, infant feeding practices, safer conception) that prevent women and men from taking full advantage of the treatment opportunities available to them and their infants. Based upon the encouraging preliminary results from our pilot study, successful CHC adoption of the "Vikela Umndeni: Protect Your Family" program could have major public health policy implications for containing the epidemic among the most vulnerable populations in rural South Africa: HIV+ pregnant women and their infants.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive pregnant women with partners, 20-24 weeks pregnant (typical time of entry into antenatal clinic care), aged >18.
* In Phase 2 (couples phase), both women and their partners will be enrolled. For the purposes of this study, primary male partners are defined as 1) husband, 2) current baby's father, or 3) current sexual partner.

Exclusion Criteria:

* Persons actively psychotic (auditory or visual hallucination) or intoxicated (e.g., under the influence of alcohol of illegal drugs) will not be eligible and will be referred for treatment. Following resolution of symptoms, these persons will be eligible for the study. N.B.: Any person presenting for sessions actively psychotic or intoxicated will be referred for treatment and will not be eligible to participate in sessions until symptoms are resolved due to reduced likelihood of benefit from sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1967 (Actual)
Dates: Start 2014-04; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Jones, PhD, Principal Investigator — University of Miami; Karl Peltzer, PhD, Principal Investigator — Human Sciences Research Council
Locations (1):
- Human Sciences Research Council, Pretoria, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Dissemination of findings will be made to the community participants and stakeholders. The US team and the South Africa team will collaborate and encourage community stakeholders to participate in dissemination and development of related research. Utilizing the data from this study, the collaborators will compile a research review document for the Government of South Africa. Successful results of this research will be used to develop a translational proposal based on empirical results. The study results will be disseminated through Dr. Peltzer, the South Africa PI. All investigators will work within the structure of the South Africa community sites to provide feedback to other medical providers and to the professional community by presentation of the results. Access to the database will be available under the supervision of the collaborators.

REFERENCES:
- [Derived] Peltzer K, Abbamonte JM, Soni M, Rodriguez VJ, Lee TK, Weiss SM, Jones DL. Psychological and physical intimate partner violence and sexual risk behavior among South African couples: a dyadic analysis. AIDS Care. 2022 Dec;34(12):1610-1618. doi: 10.1080/09540121.2021.2016576. Epub 2021 Dec 18. PMID 34927477
- [Derived] Ramlagan S, Rodriguez VJ, Peltzer K, Ruiter RAC, Jones DL, Sifunda S. Self-Reported Long-Term Antiretroviral Adherence: A Longitudinal Study Among HIV Infected Pregnant Women in Mpumalanga, South Africa. AIDS Behav. 2019 Sep;23(9):2576-2587. doi: 10.1007/s10461-019-02563-z. PMID 31228026
- [Derived] Sifunda S, Peltzer K, Rodriguez VJ, Mandell LN, Lee TK, Ramlagan S, Alcaide ML, Weiss SM, Jones DL. Impact of male partner involvement on mother-to-child transmission of HIV and HIV-free survival among HIV-exposed infants in rural South Africa: Results from a two phase randomised controlled trial. PLoS One. 2019 Jun 5;14(6):e0217467. doi: 10.1371/journal.pone.0217467. eCollection 2019. PMID 31166984
- [Derived] Peltzer K, Babayigit S, Rodriguez VJ, Jean J, Sifunda S, Jones DL. Effect of a multicomponent behavioural PMTCT cluster randomised controlled trial on HIV stigma reduction among perinatal HIV positive women in Mpumalanga province, South Africa. SAHARA J. 2018 Dec;15(1):80-88. doi: 10.1080/17290376.2018.1510787. PMID 30134772
- [Derived] Jones DL, Rodriguez VJ, Mandell LN, Lee TK, Weiss SM, Peltzer K. Influences on Exclusive Breastfeeding Among Rural HIV-Infected South African Women: A Cluster Randomized Control Trial. AIDS Behav. 2018 Sep;22(9):2966-2977. doi: 10.1007/s10461-018-2197-z. PMID 29926300
- [Derived] Peltzer K, Weiss SM, Soni M, Lee TK, Rodriguez VJ, Cook R, Alcaide ML, Setswe G, Jones DL. A cluster randomized controlled trial of lay health worker support for prevention of mother to child transmission of HIV (PMTCT) in South Africa. AIDS Res Ther. 2017 Dec 16;14(1):61. doi: 10.1186/s12981-017-0187-2. PMID 29248014
- [Derived] Jones D, Peltzer K, Weiss SM, Sifunda S, Dwane N, Ramlagan S, Cook R, Matseke G, Maduna V, Spence A. Implementing comprehensive prevention of mother-to-child transmission and HIV prevention for South African couples: study protocol for a randomized controlled trial. Trials. 2014 Oct 27;15:417. doi: 10.1186/1745-6215-15-417. PMID 25348459

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Women With Partners: Women will enroll with male partners and both members of the couple will attend the Protect your Family intervention
  Protect your family: "Protect Your Family" intervention is a manualized, closed, structured behavioral risk reduction program targeting HIV, stigma, disclosure, communication, intimate partner violence (IPV), PMTCT knowledge, safer conception, family planning and dual method sexual barrier use.
  Intervention participants will attend 3 prenatal weekly 2 hour gender-specific (male or female, 5-7 participants) group sessions followed by 1 individual counseling session and 2 monthly couples or individual (women-only) counseling sessions (1 prenatal, 2 postpartum) led by study-trained clinic staff (e.g., nurses, HIV counseling and testing (HCT) counselors) plus standard of care (PMTCT)
- Intervention Women Without Partners: Women will enroll alone and will attend the Protect your Family Intervention without a partner
  Protect your family: "Protect Your Family" intervention is a manualized, closed, structured behavioral risk reduction program targeting HIV, stigma, disclosure, communication, intimate partner violence (IPV), PMTCT knowledge, safer conception, family planning and dual method sexual barrier use.
  Intervention participants will attend 3 prenatal weekly 2 hour gender-specific (male or female, 5-7 participants) group sessions followed by 1 individual counseling session and 2 monthly couples or individual (women-only) counseling sessions (1 prenatal, 2 postpartum) led by study-trained clinic staff (e.g., nurses, HIV counseling and testing (HCT) counselors) plus standard of care (PMTCT)
Period: Overall Study
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
Started | 577 | 348 | 681 | 361
Completed | 577 | 348 | 681 | 361
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone | Total
Number analyzed (Participants) | 577 | 348 | 681 | 361 | 1967
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.24 (6.50) | 28.33 (5.58) | 30.60 (7.22) | 28.60 (5.99) | 29.73 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354 | 348 | 361 | 361 | 1424
  Male | 223 | 0 | 320 | 0 | 543
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 577 | 348 | 681 | 361 | 1967
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 577 | 348 | 681 | 361 | 1967

OUTCOME MEASURES:

1. Primary Outcome: Dried Blood Spot Analysis of Medication Adherence- Mother and Infant
Description: Presence of prescribed PMTCT protocol medications among mothers will be assessed by dried blood spot at 32 weeks gestation.
Time Frame: 32 weeks gestation
Population: The presence of medications via dried blood spot at 32 weeks gestation was only assessed in women, not infants, given that dried blood spots were not collected from infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
Number analyzed (Participants) | 67 | 204 | 54 | 242
Participants | 56 | 157 | 35 | 183
Statistical Analysis 1: Comparison: Intervention Women With Partners vs Intervention Women Without Partners vs Control Women With Partners vs Control Women Alone; Test type: Other; Odds Ratio (OR) = 1.12

2. Primary Outcome: Infant HIV Seroconversions
Description: Infants will be tested for HIV at 6 weeks per the South African standard of care and at 12 months per study protocol
Time Frame: 12 months postpartum
Population: Medical records for tests at 6 weeks were lost by the participating clinics and therefore, medical records were considered to be unreliable. Therefore, the reported results are based on 12-month tests.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
Number analyzed (Participants) | 300 | 249 | 306 | 265
Participants | 0 | 4 | 0 | 4
Statistical Analysis 1: Comparison: Intervention Women With Partners vs Intervention Women Without Partners vs Control Women With Partners vs Control Women Alone; Test type: Other; Odds Ratio (OR) = 0.32

3. Secondary Outcome: Mother Reported Rates of Infant Exclusive Breastfeeding
Description: Feeding practices will be assessed at 6 weeks, and rates of exclusive breastfeeding will be assessed.
Time Frame: 6 weeks
Population: This refers to exclusive breastfeeding as reported by the mother.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
Number analyzed (Participants) | 191 | 137 | 259 | 192
Participants | 102 | 71 | 169 | 132
Statistical Analysis 1: Comparison: Intervention Women With Partners vs Intervention Women Without Partners vs Control Women With Partners vs Control Women Alone; Test type: Other; p = 0.605, Mixed Models Analysis

4. Secondary Outcome: Attendance at Scheduled Ante and Postnatal Clinic Appointments
Description: Attendance at clinic appointments will be collected from patient records and self-report pre- and post-natal
Time Frame: 6 months postpartum
Population: Attendance records could not be retrieved for most participants. However, this analysis was still conducted among those participants who had data.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
Number analyzed (Participants) | 111 | 0 | 215 | 0
Participants | 99 | 0 | 187 |
Statistical Analysis 1: Comparison: Intervention Women With Partners vs Control Women With Partners; Attendance records could not be retrieved for most participants. However, this analysis was still conducted among those participants who had data; Test type: Other; p = 0.902, Chi-squared

5. Other Pre Specified Outcome: Self-reported Use of Condoms
Description: Sexual behavior (i.e., condom use) will be collected by participant self-report
Time Frame: 12 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
Number analyzed (Participants) | 381 | 198 | 535 | 226
Participants | 278 | 164 | 433 | 185
Statistical Analysis 1: Comparison: Intervention Women With Partners vs Intervention Women Without Partners vs Control Women With Partners vs Control Women Alone; Test type: Other; p = 0.869, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention Women With Partners vs Intervention Women Without Partners vs Control Women With Partners vs Control Women Alone; Test type: Other; p = 0.982, Mixed Models Analysis; Odds Ratio (OR) = 0.32

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored for approximately one year.
Arm/Group | Intervention Women With Partners | Intervention Women Without Partners | Control Women With Partners | Control Women Alone
All-Cause Mortality (participants affected / at risk) | 1/577 | 2/348 | 0/681 | 1/361
Serious Adverse Events (participants affected / at risk) | 0/577 | 0/348 | 0/681 | 0/361
Other Adverse Events (participants affected / at risk) | 0/577 | 0/348 | 0/681 | 0/361

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02085356/Prot_SAP_000.pdf